CLINICAL TRIAL: NCT02740621
Title: Evaluation of Past Medications in Patients With Coronary Heart Disease and Patients Hospitalized for a Non-cardiac Reason
Brief Title: The Impact of Opioids in Coronary Heart Disease
Acronym: MIOP/TRAPS
Status: Completed | Type: Observational
Sponsor: Ruhr University of Bochum (Other)
Collaborators: Mundipharma Research GmbH & Co KG (Industry)
Responsible Party: Principal Investigator, Christoph Maier, Prof. Dr., Prof., Dr., Ruhr University of Bochum
Other Study IDs: MIOP
Record Dates: First submitted 2016-03-30; First posted 2016-04-15 (Estimated); Last update posted 2018-04-11 (Actual); Status verified 2018-04

CONDITIONS: Coronary Heart Disease
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with coronary heart disease: coronary angiography with finding coronary heart disease currently no cancer 40 years or older
- control patients: coronary angiography with exclusion coronary heart disease or other patients with non-cardiac diseases currently no cancer 40 years or older

SUMMARY:
In this study, the risk of opioid medications on coronary heart disease in adults is investigated. Patients with the necessity of a coronary angiography and control patients with a non-cardiac disease of the same hospital are inquired with a standardized questionnaire about demographic and clinical risk factors for heart attack. An impact of opioid medications on coronary heart disease is hypothesised (MIOP).

In addition, all patients with coronary angiography should be consulted twice (after 3 and 6 months) to find out how many of these patients have developed a refractory angina pectoris (TRAPS).

ELIGIBILITY:
Inclusion Criteria:

* 40 years or older
* written informed consent

Exclusion Criteria:

* currently cancer
* cognitive limitations

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: hospitalized patients in University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 750 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Number of patients with opioid treatment (WHO II/ WHO III) within the last 10 years before present hospitalization, Interview with standardized CRF | 20 minutes
  Standardized assessment of opioid medications taken before hospital admission to evaluate the impact of opioids in coronary heart disease.
  Exact doses, substances and intake habits are inquired.
Number of patients with refractory angina pectoris, Interview with standardized CRF | 30 minutes
  Standardized assessment of angina pectoris symptoms and treatments to evaluate a refractory angina pectoris.
  Changes of their medications are inquired twice.

CONTACTS AND LOCATIONS:
Locations (1):
- Bergmannsheil department of pain therapy, Bochum, North Rhine-Westphalia, Germany